CLINICAL TRIAL: NCT02016989
Title: REGENERATING AGENT (OTR4120) AND BACTERIAL KERATITIS : A RANDOMISED TRIAL
Brief Title: Matrix Therapy And Bacterial Keratitis
Acronym: CACICOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0169; 2013-A01166-39
Record Dates: First submitted 2013-11-25; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Bacterial Keratitis
Keywords: Bacterial keratitis; OTR4120; Matrix therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Physiological salt solution (Other): The purpose of this study is to evaluate efficiency of CACICOL20 for bacterial keratitis. It is a double blinded comparison of epithelial defect in two groups of patients randomized between CACICOL20 and physiological salt solution.
  Interventions: Device: physiological salt solution
- CACICOL20 (Experimental): The purpose of this study is to evaluate efficiency of CACICOL20 for bacterial keratitis. It is a double blinded comparison of epithelial defect in two groups of patients randomized between CACICOL20 and physiological salt solution.
  Interventions: Device: RGTA OTR4120 (CACICOL20)

INTERVENTIONS:
Device: RGTA OTR4120 (CACICOL20)
  Arms: CACICOL20
Device: physiological salt solution
  Arms: Physiological salt solution

SUMMARY:
The purpose of this study is to evaluate efficiency of CACICOL20 for bacterial keratitis. It is a double blinded comparison of epithelial defect in two groups of patients randomized between CACICOL20 and physiological salt solution.

DETAILED DESCRIPTION:
Extracellular matrix, composed of glycosaminoglycans (GAG) and matricial proteins, has a key role in tissular homeostasis.

The matrix therapy is a new class of medical substance, called RGTAs, ReGeneraTing Agents, consist of chemically engineered polymers adapted to interact with and protect against proteolytic degradation of cytokines.

OTR4120 (CACICOL20) is an heparan sulphate (HS) mimetic that can replace the degraded HS and protect and improve the bioavailability of cytokines. It aims to facilitate and potentiate the wound healing by restorating the natural microenvironment.

CACICOL20 was used in treating corneal dystrophies and chronic corneal ulcers. It significantly favored corneal healing. It was well tolerated with no side effects.

Bacterial keratitis is a serious ocular condition that may result in significant sight-threatening corneal sequelae. The common risk factors for infectious keratitis include ocular trauma, contact lens wear, recent ocular surgery, preexisting ocular surface disease, dry eyes, lid deformity, corneal sensational impairment, chronic use of topical steroids, and systemic immunosuppression. Serious cases of keratitis are hospitalized to administrate an intensive hospital-made local antibiotic.

The purpose of this study is to evaluate efficiency of CACICOL20 for bacterial keratitis. It is a double blinded comparison of epithelial defect in two groups of patients randomized between CACICOL20 and physiological salt solution.

ELIGIBILITY:
Inclusion Criteria:

* - Hospitalized patients for bacterial keratitis in Ophthalmology Department, Clermont-Ferrand university hospital .with a controlled local infection after 48 hours local antibiotics.

  * with a corneal ulcer diameter > 2 millimeters

Exclusion Criteria:

* - Ulcers deeper than the superficial stroma, perforated ulcers or pre-perforated, requiring a surgical intervention < 15 days.
* Clinical suspicion and/or microbiological evidence of fungal or parasitic infection
* Non controlled infection in spite of 48 hours intensive local antibiotics
* Allergy
* Silver or copper salts treatment
* Ocular surgery within the last 1 month
* Unable to follow up medical examinations for geographical, social, physical or psychological reasons
* Patient already included in another clinical trial
* Pregnant patients or breastfeeding
* Person under a legal protection measure, under guardianship
* Not cover by social insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Epithelial corneal surface healing | at day 1
  each day, from date of randomization until the date of the complete corneal healing assessed to fifteen days, up to 2 months

SECONDARY OUTCOMES:
Healing time of total corneal epithelial wound | at day 1
  each day, from date of randomization until the date of the complete corneal healing assessed to fifteen days, up to 2 months
Visual acuity | at day 1 and day 12
  date of randomization and date of the complete corneal healing
Ulcer deep | every day between day 0 to day 12
  every two days, from date of randomization until the date of the complete corneal healing assessed to fifteen days, up to 2 months
Healing keratitis rate | at day 12
  at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric CHIAMBARETTA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France